CLINICAL TRIAL: NCT00003748
Title: Phase II Study of Irinotecan (CPT-11) in Adenocarcinoma of the Esophagus and Gastric Cardia
Brief Title: Irinotecan in Treating Patients With Esophageal or Stomach Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: Pharmacia and Upjohn (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066868; UCLA-HSPC-9703008; P-UPHJOHN-6475-96014; NCI-G99-1497
Record Dates: First submitted 1999-11-01; First posted 2004-07-22 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2012-07

CONDITIONS: Esophageal Cancer; Gastric Cancer
Keywords: stage I gastric cancer; stage II gastric cancer; stage III gastric cancer; stage IV gastric cancer; recurrent gastric cancer; stage I esophageal cancer; stage II esophageal cancer; stage III esophageal cancer; stage IV esophageal cancer; recurrent esophageal cancer; adenocarcinoma of the stomach; adenocarcinoma of the esophagus
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms; Adenocarcinoma Of Esophagus | interventions — Irinotecan

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- irinotecan hydrochloride (Experimental): One course of therapy is comprised of a 4-week treatment period and a two-week rest period. Drug administration will be based on actual calculated body surface area. Starting dose will be 125 mg/m2/day given once per week on four consecutive weeks.
  Interventions: Drug: irinotecan hydrochloride

INTERVENTIONS:
Drug: irinotecan hydrochloride — One course of therapy is comprised of a 4-week treatment period and a two-week rest period. Drug administration will be based on actual calculated body surface area. Starting dose will be 125 mg/m2/day given once per week on four consecutive weeks.
  Other Names: CPT-11

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die.

PURPOSE: Phase II trial to study the effectiveness of irinotecan in treating patients who have esophageal or stomach cancer.

DETAILED DESCRIPTION:
OBJECTIVES: I. Determine the antitumor activity of irinotecan in patients with adenocarcinoma of the esophagus or gastric cardia. II. Evaluate the toxicities of this drug in this patient population.

OUTLINE: This is a multicenter study. Patients receive irinotecan intravenous (IV) over 90 minutes once a week for 4 weeks followed by a 2 week rest period. Treatment continues in the absence of unacceptable toxicity or disease progression. Patients are followed every 3 months until death.

PROJECTED ACCRUAL: A total of 18-32 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Patients must be > 18 years of age
* Patients must have a performance status of 0-2 on the Eastern Cooperative Oncology Group (ECOG) Performance Scale
* Patients must have a predicted life expectancy of at least 12 weeks
* Patients must have a pretreatment granulocyte count of >1500/mm3, a hemoglobin level of >9.0 gm/dL and the platelet count of >100000/mm3
* Patients must have adequate renal function as documented by a serum creatinine < 2.0 mg/dL
* Patients must have adequate hepatic function as documented by a serum bilirubin < 1.5 mg/dL, regardless of whether patients have liver involvement secondary to tumor. Aspartate transaminase must be < 3 x institutional upper limit of normal unless the liver is involved with tumor, in which case the aspartate transaminase must be < 5 x institutional upper limit of normal
* Patients must have histologically proven adenocarcinoma of the esophagus or gastric cardia with progression despite prior chemotherapy
* Patients must have disease radiologically measurable bidimensionally
* Patients must have an interval of 4 weeks from prior chemotherapy, immunotherapy, or radiation therapy

Exclusion Criteria:

* Patients with any active or uncontrolled infection
* Patients with psychiatric disorders that would interfere with consent or follow-up
* Patients with a history of myocardial infarction within the previous six months or congestive heart failure requiring therapy
* Patients with a history of prior malignancy except for adequately treated basal cell or squamous cell skin cancer, in situ cervical cancer, or other cancer for which the patient has been disease-free for at least five years
* Pregnant or lactating women. Men and women of reproductive potential may not participate unless they have agreed to use an effective contraceptive method
* Presence of clinically apparent central nervous system metastases or carcinomatous meningitis
* Patients with uncontrolled diabetes mellitus
* Patients with any other severe concurrent disease which, in the judgment of the investigator, would make the patient inappropriate for entry into this study
* Prior therapy with a deoxyribonucleic acid (DNA) topoisomerase inhibitor
* Patients with known Gilbert's syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 1998-08; Primary Completion 2000-06 (Actual); Study Completion 2005-01 (Actual)

PRIMARY OUTCOMES:
To determine the antitumor activity of irinotecan hydrochloride (CPT-11) in patients with unresectable adenocarcinoma of the esophagus and gastric cardia who have failed prior chemotherapy | 2 years

SECONDARY OUTCOMES:
Evaluate the toxicities of irinotecan hydrochloride (CPT-11) in the patient population | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Joel R. Hecht, MD, Principal Investigator — Jonsson Comprehensive Cancer Center
Locations (25):
- United States (25):
  - Comprehensive Blood and Cancer Center, Bakersfield, California
  - St Jude Heritage Health Foundation, Fullerton, California
  - Daniel Freeman Memorial Hospital, Inglewood, California
  - UCLA - Antelope Valley Cancer Center, Lancaster, California
  - Pacific Shores Medical Group, Long Beach, California
  - Jonsson Comprehensive Cancer Center, UCLA, Los Angeles, California
  - Community Hospital of the Monterey Peninsula, Monterey, California
  - Office of Jerome L. Rubin, Monterey, California
  - Office of Eddie Hu, M.D., Monterey Park, California
  - Ventura County Hematology-Oncology Medical Group, Inc., Oxnard, California
  - Wilshire Oncology Medical Center, Pomona, California
  - Salinas Valley Memorial Hospital, Salinas, California
  - Cancer Center of Santa Barbara, Santa Barbara, California
  - Sansum Medical Clinic, Santa Barbara, California
  - James L. Poth, M.D., Michael Alexander, M.D., Inc., Santa Cruz, California
  - Marian Medical Center, Santa Maria, California
  - Office of Marilou Terpenning, Santa Monica, California
  - Office of Robert C. Klein, Santa Monica, California
  - Dominican and Watsonville Community Hospital, Soquel, California
  - Los Robles Regional Medical Center, Thousand Oaks, California
  - Cancer Care Associates Medical Group, Torrance, California
  - UCLA Cancer Center - Santa Clarita, Valencia, California
  - Oncology Medical Center of North County, Vista, California
  - Valley Hematology and Oncology, West Hills, California
  - Cancer Care Consultants, Las Vegas, Nevada